CLINICAL TRIAL: NCT02642939
Title: A Phase II Study of Treatment With Oral Mifepristone as Salvage Therapy in Patients With Advanced or Metastatic Non-Small Cell Lung Cancer Who Have Failed Two or More Previous Chemotherapy Regimens
Brief Title: Study of Oral Mifepristone as Salvage Therapy in Patients With Advanced or Metastatic Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Check, Jerome H., M.D., Ph.D. (Individual)
Collaborators: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIF-01-2014
Record Dates: First submitted 2015-12-11; First posted 2015-12-30 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Mifepristone; Corlux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- mifepristone (Experimental): mifepristone 300 mg capsule per day, orally in 28-day cycles
  Interventions: Drug: Mifepristone

INTERVENTIONS:
Drug: Mifepristone — Mifepristone is an antagonist of the GR-II (glucocorticoid) receptor, yet has little affinity for the GR-I (mineralocorticoid) receptor. Mifepristone is also a potent antagonist at the progesterone receptor, and may block the androgen receptor to a limited degree.
  Other Names: KORLYM®, C1073, CORLUXIN™ and CORLUX™.

SUMMARY:
This is a non-randomized, multicenter, single-stage phase II study of mifepristone in patients with advanced or metastatic NSCLC who have failed two or more previous chemotherapy regimens.

The Investigator plans to enroll 18 evaluable patients in Stage 1, and additionally up to 22 evaluable patients in Stage 2 for a total of 40 evaluable patients. Participants will be followed for overall survival. Current salvage therapy in advanced NSCLC achieves a median progression free survival time of 10 weeks and overall survival of 10 months. The Investigator would like to provide evidence that mifepristone will increase the median progression-free survival time to 15 weeks and overall survival time of 16 months.

DETAILED DESCRIPTION:
This is a non-randomized, multicenter, single-stage phase II study of mifepristone in patients with Stage IIIB or Stage IV NSCLC who have failed two or more previous chemotherapy regimens.

The primary objective of this trial is to evaluate the utility of mifepristone as a salvage therapy in patients with Stage IIIB or Stage IV non-small cell lung carcinoma who have failed at least two previous chemotherapy regimens. Efficacy will be measured by improvement in progression-free survival and life span; and overall response as compared to historical controls.

Plan to enroll 18 evaluable patients in Stage 1 and up to 22 evaluable patients in Stage 2 for a total of 40 evaluable patients. Anticipated duration of the study is approximately up to 36 months.

Patients who tolerate treatment in the first cycle are eligible to continue to receive treatment until they experience unacceptable toxicity, until they meet any of the withdrawal criteria, or until the study is terminated by the Sponsor.

Patient may continue treatment despite evidence of tumor progression if they feel better, i.e. improved quality of life.We will follow all patients for overall survival.

Current salvage therapy in advanced NSCLC achieves a median progression free survival time of 10 weeks and overall survival of 10 months. We would like to provide evidence that mifepristone will increase the median progression-free survival time to 15 weeks and overall survival time of 16 months.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet the following criteria to be enrolled in the study

1. Must understand and voluntarily sign an informed consent
2. Age ≥ 18 years at the time of signing the informed consent
3. Histological or cytological documented diagnosis of locally advanced, recurrent or metastatic (Stage IIIB or Stage IV) NSCLC
4. Patients must have evidence of disease, measurable or evaluable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST v1.1).
5. Patients shall provide results of tumor testing for epidermal growth factor receptor (EGFR) mutation or anaplastic lymphoma kinase (ALK) rearrangement, and if positive for EGFR mutation or ALK rearrangement shall have received appropriate targeted therapy prior to enrollment. If not previously tested, EGFR and ALK testing must be performed prior to study entry.
6. Patients shall have progressed after two or more previous chemotherapy regimens for metastatic or locally advanced disease
7. Patients must have recovered from any toxic effects and at least 3-4 weeks must have elapsed from the last dose of previous therapy, prior to registration
8. Eastern Cooperative Oncology Group (ECOG) performance status 0 - 3
9. Life expectancy of at least 12 weeks
10. Patients must have adequate bone marrow and renal/hepatic function at the screening visit, defined as:

    * Absolute neutrophil count ≥ 1,500/mm3 without granulocyte colony-stimulating factor (G-CSF) support within 7 days preceding the lab assessment
    * Platelet count ≥ 100,000/mm3, without transfusion within 7 days preceding the lab assessment
    * Hemoglobin ≥ 9 g/dL, without transfusion support within 7 days preceding the lab assessment
    * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 3 × upper limit of normal (ULN)
    * Total serum bilirubin ≤ 1.5 times ULN
    * Serum creatinine ≤ ULN
    * Potassium and magnesium levels within normal limits. Patients with potassium or magnesium below the lower limit of normal must have levels corrected to normal by supplementation prior to starting study drug
11. Disease-free period of > 3 years from any other previous malignancies, excluding curatively treated basal cell carcinoma, squamous cell carcinoma of the skin, or carcinoma in situ of the cervix
12. Female patient of childbearing potential must have a negative serum pregnancy test. Sexually active female patient f childbearing potential must be willing to use non-hormonal contraception, including condom use by male partner, and barrier method by the female partner (diaphragm or cervical cap both with spermicide) during the treatment period and for at least 3 months after the last dose of the study drug. Females considered not of childbearing potential include those who have been in menopause at least 2 years, or are surgically sterile (status post tubal ligation or hysterectomy).
13. Patients must be able and willing to comply with the study visit schedule and study procedures
14. Able to take oral medications.

Exclusion Criteria:

Patients who meet any of the following criteria will not be permitted entry to the study:

1. Pregnant or breast-feeding
2. Women with a history of unexplained vaginal bleeding.
3. Women with uterine hyperplasia - in pre-menopausal women hyperplasia >18mm and in post-menopausal women hyperplasia of >10mm Prior therapy with mifepristone
4. Prior therapy with mifepristone
5. Patients who have had recent systemic cytotoxic therapies or radiotherapy within 14 days prior to day 1 of cycle 1
6. Use of cytotoxic chemotherapeutic agents, erythropoiesis-stimulating agents (ESA), or experimental agents (agents that are not commercially available) within 30 days of the first day of study drug treatment.
7. Patients who have had any major surgery within 4 weeks prior to day 1 of cycle 1, or minor surgery within 2 weeks prior to day 1 of cycle 1
8. For two weeks prior to first day of study drug treatment, administration of any of the following cytochrome P450 3A (CYP3A) inducers: phenytoin, phenobarbital, carbamazepine, rifampin, rifabutin, St. John's Wort; or CYP3A inhibitors: ketoconazole, itraconazole, nefazodone, ritonavir, nelfinavir, indinavir, atazanavir amprenavir, fosamprenavir, boceprevir, clarithromycin, conivaptan, lopinavir, posaconazole, saquinavir, telaprevir, telithromycin, or voriconazole
9. Patients who are taking simvastatin or lovastatin. Patients should be switched to alternative therapies a minimum of 2 weeks before starting study drug
10. Patients who have been treated with an investigational agent within 21 days prior to day 1 of cycle 1.
11. Concomitant use of biological agents including growth factors
12. Patients who require treatment with systemic corticosteroids for serious medical conditions or illnesses (e.g. immunosuppression after organ transplantation)
13. Chronic liver disease as indicated by Child-Pugh score A (6) or greater
14. History of significant cardiac disease. Significant cardiac diseases includes second/third degree heart block; significant ischemic heart disease; mean QTc interval > 480 msec on at least two separate electrocardiograms (ECGs) prior to study start; poorly controlled hypertension; congestive heart failure of New York Heart Association (NYHA) Class II or worse (slight limitation of physical activity; comfortable at rest, but ordinary physical activity results in fatigue, palpitation, or dyspnea)
15. Any other significant co-morbid conditions that in the opinion of the investigator would impair study participation or cooperation
16. Concomitant use of progestational agents
17. Known history of human immunodeficiency virus (HIV) positivity
18. In the opinion of the Investigator, any serious medical condition or psychiatric illness that will prevent the patient from signing the informed consent or will place the patient at unacceptable risk if he/she participates in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Overall Survival | through study completion, an average of 16 months
  defined as the time from first dose of study drug to the date of death
A. Improvement in Quality of Life (QoL) | every 8 weeks from date of enrollment until end of study or the date of death from any cause, assessed using QoL questionnaire,assessed up to 56 months.
  Participants complete QoL questionnaire EROTC QLQ-C30 every 8 weeks
B. Improvement in Quality of Life (QoL) | every 8 weeks from date of enrollment until end of study or the date of death from any cause, assessed using QoL questionnaire,assessed up to 56 months.
  Participants complete QoL questionnaire EROTC QLQ-LC13 (specific to lung cancer)

SECONDARY OUTCOMES:
Progression free survival | median of 15 weeks from study enrollment until end of study or the date of first documented progression, assessed every 12 weeks by radiologic examination,assessed up to 56 months.
  defined as the time from first dose of study drug to the date of the first documented tumor progression (per RECIST 1.1) or death due to any cause
Overall response rate | assessed every 4 weeks, from date of enrollment until end of study or the date of death from any cause, assessed up to 56 months.
  defined as the number of subjects whose best confirmed objective response is either a complete response (CR) or partial response (PR) divided by the number of randomized subjects
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | assessed every week for 1 month and then every 4 weeks, from date of enrollment until end of study or the date of death from any cause, assessed up to 56 months.
  to determine any toxicity from the drug at the 300 mg dosage.

CONTACTS AND LOCATIONS:
Overall Officials: Jerome H Check, MD,PhD, Principal Investigator — Cooper Institute for Reproductive Hormonal Disorders
Locations (1):
- Cooper Institute for Reproductive Hormonal Disorders, Melrose Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
See below
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 1 year after completion of study